CLINICAL TRIAL: NCT06717256
Title: Evaluation of the Effect of Nurse Coaching Program on Self-management and Skin Care Behaviors in Patients With Diabetes: a Randomized Controlled Trial.
Brief Title: Evaluation of the Effect of Nurse Coaching Program on Self-management and Skin Care Behaviors in Patients With Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Burcu Kuccuk, Student, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NecmettinEU-SBF-BK-01
Record Dates: First submitted 2024-12-01; First posted 2024-12-04 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus Self Management Education; Diabetes Mellitus, Type II; Skin Care
Keywords: Diabetes Mellitus Self Management Education; Skin Care; Tip II Diyabet Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Self-Management

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EDUCATION GROUP (Experimental): In addition to routine training provided by physicians to patients in this group, training will be provided within the first 6 weeks, where "the effect of the nurse coaching program on self-management and skin care behaviors in diabetic patients will be evaluated" and monthly reminders will be provided thereafter. The content of the training booklet prepared for self-management and skin care will be presented to the participants as a face-to-face training in the form of one-week presentations to be completed in 6 weeks, in the form of oral presentations. At the end of the module training, participants will be asked questions and answered. Six weeks after the training is completed, participants will be provided with reminders, and the trainings they want to be repeated will be repeated.
  Interventions: Behavioral: training
- CONTROL GROUP (No Intervention): Participants assigned to the control group will receive information training as part of their check-ups, as in routine practice; however, the intervention program evaluating the effect of the nurse coaching program on self-management and skin care behaviors in diabetic patients will not be implemented.

INTERVENTIONS:
Behavioral: training — The diabetes education booklet is a collection of information designed by the researcher. These interventions will continue for 1.5 months, with a total of 6 sessions for each type 2 DM individual, lasting approximately 120 minutes (2 hours per week and 12 hours in total after 6 weeks), and will be carried out as reminders afterwards. In these sessions, agendas will be created appropriately on regular eating habits, physical activity, regular monitoring of blood sugar, compliance with treatment, problem-solving ability, coping strategies and minimizing risks, conflicts regarding self-management and skin care behaviors of the patient will be tried to be resolved, the patient's suitability and adaptation to the change phase will be determined, their willingness to change will be questioned, and the change plan will be helped in the matters of care and self-management.
  Other Names: scin care; self-management
  Arms: EDUCATION GROUP

SUMMARY:
This research will be conducted in a pre-test-post-test randomized controlled, single-blind experimental design to evaluate the effects of a nurse coaching program on self-management and skin care behaviors in patients with diabetes. The key question(s) it aims to answer are:

* Does the nurse coaching program have no effect on self-management behaviors and skin care behaviors in patients with diabetes?
* Does the nurse coaching program have no effect on self-management behaviors and skin care behaviors in patients with diabetes?

DETAILED DESCRIPTION:
The study will be conducted in the internal medicine units of Mut State Hospital in the Mut district of Mersin between January 2025 and June 2025. An average of 100 patients with type 2 DM apply to the hospital per day. According to Cohen's effect size coefficients; it was decided to include 21 people (N=42) in the groups, assuming that the evaluations to be made between two independent groups would have a large effect size (d=0.8; large) according to the calculations made. The consents of 42 type 2 DM patients who constitute the study group of the experimental research will be obtained. After the preliminary tests are performed, a series of random numbers will be generated by an independent statistician and 21 will be assigned to the intervention group and 21 to the control group using the simple randomization method.

Personal Information Form, Diabetes Self-Management Scale, and Skin Care Behavior Monitoring Form will be used as Data Collection Tools. In addition, the "Diabetes Education Booklet" designed and prepared by the researchers will be used as an intervention material in the research study.The follow-up of the implementation process will be recorded with the MSF and KBIF prepared by the researcher.Before starting the research, 3 measurements will be taken at week 6 and week 12. The data collection process of the research will be completed by using face-to-face training opportunities in the first 6 weeks and reminders (message, phone call, etc.) in the following periods. The control group will receive standard training and the same measurement tools will be used.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65,
* Having a Type 2 DM diagnosis period of 6 months or more,
* Not having any psychiatric disorders or mental problems,
* Having hemoglobin A1c values <8 mmol/mL,
* Individuals who can perform diabetes self-management behaviors and skin care behaviors (regular eating habits, physical activity, regular monitoring of blood sugar, compliance with treatment, ability to solve problems, coping strategies and minimizing risks).

Exclusion Criteria:

* Exclusion criteria for the study;
* Having verbal communication problems,
* Having been diagnosed with Type 1 Diabetes Mellitus,
* Having been diagnosed with gestational diabetes mellitus,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
PERSONAL INFORMATION FORM | Before the study.
  A two-part personal information form prepared by the researcher based on the literature (Herath et al. 2017; Kassahun et al. 2017; Ahmed et al. 2019; ADA 2021; Alaofè et al. 2021) was used. The Personal Information Form consists of 7 questions about socio-demographic characteristics (age, gender, marital status, educational status, presence of health insurance, economic status, place of residence) and 7 questions about disease-health characteristics (blood sugar measurement status, ability to take medications regularly, presence of any chronic disease other than diabetes, status of consulting a doctor for diabetes control, exercise status, status of receiving sufficient education regarding diabetes, if the answer is yes, what trainings have been received, measured HbA1C result).

SECONDARY OUTCOMES:
Diabetes Self Management Questionnaire | Before application, at week 6 of application and at week 12 of application
  This scale is a 16-item individual assessment scale developed by Schmitt et al. in 2013 to examine the relationship between diabetes self-management and glycemic control in diabetic patients. Participants are asked to answer the questions by considering their condition in the last 8 weeks. In the validity and reliability study conducted with 261 diabetic patients, Cronbach's alpha value was found to be 0.84. In the validity and reliability study conducted by Eroğlu and Sabuncu (2018), Cronbach's alpha value was found to be 0.85. The scale consists of 4 sub-dimensions. --Glucose Management: 1, 4, 6, 10, 12 (items 4 and 12 are related to medication use, items 1, 6 and 10 are related to blood sugar monitoring)
  * Diet Control: 2, 5, 9, 13
  * Physical Activity: 8, 11, 15
  * Health Services Use: 3, 7, 14 Item 16 is not included in any sub-dimension. The scale is a 4-point Likert type.

OTHER OUTCOMES:
Skin Care Behavior Monitoring Form | before application, at week 6 of application and at week 12 of application
  It consists of 20 questions that will evaluate the general skin care practices of individuals with type 2 DM. All questions will be positive. Individuals with positive general skin care behaviors are expected to mark "yes" to all questions. Participants will answer the questions as "yes" and "no". The number of "yes" answers of individuals with type 2 DM regarding general skin care behaviors will be taken into account in the evaluation of the form. In order to evaluate the general skin care behavior status of individuals as good, they must mark yes to all 20 questions specified in the form. Those who mark 10 questions and below as "yes" in the form will be evaluated as having poor general skin care behavior status.

IPD SHARING:
Plan to Share IPD: No